CLINICAL TRIAL: NCT05896995
Title: Investigation of the Efficiency of Different Exercise Approaches in Individuals Providing Primary Care to Multiple Sclerosis Patients
Brief Title: Efficiency of Different Exercise Approaches in Individuals Providing Primary Care to MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-07/02
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Back Pain
Keywords: back pain; multiple sclerosis
MeSH Terms: conditions — Back Pain; Multiple Sclerosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Exercise (Experimental): pilates exercise+ Mckenzie Exercise Six weeks, twice a week
  Interventions: Other: Pilates Exercise
- Mckenzie Exercise (Active Comparator): Mckenzie Exercise Six weeks, twice a week
  Interventions: Other: Mckenzie Exercise

INTERVENTIONS:
Other: Pilates Exercise — Pilates exercises target the deep muscles of the core, including the abdomen, lower back, hips, and glutes, while also engaging the whole body.
  Arms: Pilates Exercise
Other: Mckenzie Exercise — The McKenzie Method emphasizes self-treatment and active patient involvement in the management of their condition. It involves a systematic assessment process to determine the most appropriate exercises and interventions for an individual based on their specific symptoms and movement responses.
  Arms: Mckenzie Exercise

SUMMARY:
Multiple Sclerosis is known as an inflammatory central nervous system disease characterized by demyelination and axonal damage.

DETAILED DESCRIPTION:
Individuals with MS cannot perform self-care in many areas due to the problems they encounter during their daily life activities, and they need an individual who will take care of them and a lifelong care.

ELIGIBILITY:
Inclusion Criteria

* Chronic low back pain he is 18-60 years old
* No verbal communication barrier
* Complaining of pain for more than three months
* Volunteering of participants Exclusion Criteria
* Absence of cognitive impairment (delirium, dementia, amnesia)
* Exercise contraindications (uncontrolled medical conditions)
* Caring for individuals with an unclear diagnosis of MS
* Disagreeing with the measurements to be made or providing incomplete answers
* Previous spinal surgery
* Spinal and joint disorders other than lumbar disc herniation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 6 weeks
  It is a questionnaire to evaluate the disability levels and quality of life faced by patients due to low back pain. It was developed to evaluate pain-related limitation in people with acute, subacute, or chronic low back pain. It includes 1 item related to pain and 9 items related to activities of daily living (personal care, lifting, walking, sitting, sanding, sleep, sexual life, social life and travel). Each item is measured on a 6-point rank scale between 0 and 5 points according to the scenarios it contains. At the end of the survey, the scores are summed and the percentage value is calculated for the total score.
Beck Depression Scale | 6 weeks
  This scale has been shown to accurately measure the level of depression. The scale consists of 21 questions with 4 options, each corresponding to 0-3 points, and the patient is asked to choose the appropriate sentence according to his condition in the last week. mood, pessimism, sense of failure, dissatisfaction, sense of guilt, sense of punishment, self-hatred, self-blame, desire for self-punishment, crying spells, irritability, social introversion, indecisiveness, deterioration of body perception, determination of workability, sleep disorders, 21 symptoms and behaviors including fatigue, fatigue, decreased appetite, weight loss, somatic complaints and loss of libido are questioned.
Bakas Caregiver Impact Scale. | 6 weeks
  It evaluates the opportunity and power of caregiving for caregivers. The scale includes a total of 15 questions scored between +3 (best aspect) and -3 (worst aspect). It is a Likert-type scale with questions from 1 to 7 according to the answers that are affected by creation or negative effects. The worst affected person can get 15 points and the best affected person can get 105 points. As the score rises, it takes shape as "good influence", and as the score decreases, it takes shape as "bad influence".
Disability status assessment. | 6 weeks
  A single EDSS score between 0-10 is determined according to the scores obtained from the functional systems. While 0 points on the scale indicate normality, 10 points indicate the way of death when MS is sufficient. In the scale, the first score that can be obtained after 0 is 1. It is a beloved scale to see if there is an index in case of disability.
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | 6 weeks
  It consists of 54 items, 2 main groups, 12 subgroups and 2 independent items: body organs health and places mental health (BMS). BFS units are in 8 subgroups: physical health, limitation due to physical devices, pain sensation, fatigue, social functionality, health perception, health distress, sexual functionality. BFS and BMS scores, which are the two main groups of the MSQOL-54 scale, are scored between 0-100. The high score obtained from the scale determines the goodness of life quality.
Algometer | 6 weeks
  An objective method, a manual algometer device, was used to assess pain sensitivity to pressure. In this study, "Baseline Dolorimeter" was preferred. The measurement was aimed at the unilateral iliocostalis lumborum muscle. Individuals were asked to say as soon as the feeling of pressure turned into a feeling of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No